CLINICAL TRIAL: NCT05384483
Title: Vraylar® (Cariprazine) in the Treatment of Social Anxiety Disorder: A Double-Blind Study
Brief Title: Cariprazine Versus Placebo for Social Anxiety Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Medical Research Network (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VRA-MRN-S40
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Social Anxiety Disorder
Keywords: SAD; Social Anxiety; Social Phobia; Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social | interventions — cariprazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cariprazine (Experimental): Cariprazine 1.5 to 3 mg per day
  Interventions: Drug: Cariprazine
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cariprazine — Cariprazine 1.5 to 3 mg per day
  Other Names: Vraylar®
  Arms: Cariprazine
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
The proposed study is a 12 week double-blind, placebo-controlled trial to examine the efficacy, safety, and tolerability of Vraylar® (cariprazine) in the treatment of patients with Social Anxiety Disorder (SAD), as defined by the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5). Subjects will be randomized to one of two treatment arms (placebo or Vraylar® 1.5 mg/day) in a 1:1 ratio. The study will be done at a single clinical research site.

DETAILED DESCRIPTION:
Social Anxiety Disorder is recognized as a prevalent, chronic and disabling condition (Schneier et al, 1992). Lifetime prevalence has been estimated at 13% in the National Comorbidity Survey (NCS (Magee et al, 1996)). The age of onset of Social Anxiety Disorder (SAD) is early, usually in the teenage years, and social, academic and vocational impairment are often severe (Schneier et al, 1992; Stein et al, 2000). Depression and alcohol abuse are common sequelae.

There is a need for more therapeutic agents for Social Anxiety Disorder. At this time, only Paxil (paroxetine), Zoloft (sertraline), Luvox CR (fluvoxamine maleate), and Effexor XR (venlafaxine) are approved. However, each of these agents helps only about 45-55% of a given sample. Furthermore, the majority of those considered responders after an acute trial are still clinically symptomatic. The same can be said for the most effective form of psychosocial treatment for social anxiety disorder, Cognitive Behavior Therapy (CBT) (Heimberg et al, 1998), and other effective drug treatments such as phenelzine (Liebowitz et al, 1992) and clonazepam (Davidson et al, 1993). In addition, all of the drug treatments found effective to date have troubling adverse effects such as weight gain, sexual dysfunction, physical dependency, or inducing tolerance that can make long term use difficult. Thus, additional treatments are needed for Social Anxiety Disorder.

Vraylar® should be helpful for patients with SAD. It is a partial agonist at D2 and D3 receptors with affinity as well for a variety of serotonin receptors including 5-HT1A, 5-HT 2A 5-HT 2C and 5-HT 7. While it has been most extensively studied for its antipsychotic and anti-manic properties, its serotonergic and dopaminergic receptor profile suggests it may also be helpful for anxiety states. Social Anxiety Disorder is an excellent area to assess a medication's anti-anxiety properties. The disorder's high prevalence makes study enrollment fairly straightforward. Its chronicity mitigates against placebo response, which has been in the 30% range in most placebo-controlled trials. The most commonly used rating instrument for SAD, the Liebowitz Social Anxiety Scale (LSAS), has demonstrated validity and reliability. Most striking is the consistency and reproducibility of results from one trial to the next with the same agent. Registration trials for Zoloft® were 2 for 2 positive, for Paxil® 3 for 3, and for Effexor® XR 5 for 5. Finally, medications found effective for SAD have also been shown to work in generalized anxiety disorder, suggesting SAD as a good indication for proof of concept studies to test a medication's antianxiety properties.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults between 18 and 65 years of age (inclusive).
* Subjects must give written informed consent prior to any study procedures.
* Diagnosis of Social Anxiety Disorder (SAD) (300.23 Social Anxiety Disorder) according to DSM-5 criteria, as determined by psychiatric evaluation with the Investigator and confirmed by the Mini-International Neuropsychiatric Interview (MINI).
* Subjects must have a minimum total score of 70 on the LSAS at both Screening and Baseline visits.
* Subjects must have a total Hamilton Depression Rating Scale (HAM-D) score of less than 16 at the Screening and Baseline visits.
* Subjects must have a Clinical Global Impression of Severity (CGI-S) score of 4 or greater at both Screening and Baseline visits.
* All subjects of childbearing potential must commit to an effective form of contraception for the duration of the trial and for at least 4 weeks after it ends. Effective forms of contraception include: condoms with spermicide, diaphragm with spermicide, hormonal contraceptive agents (oral, transdermal, or injectable), or implantable contraceptive devices. Abstinence from heterosexual intercourse will also be considered an effective form of contraception, if abstinence is part of the subject's usual lifestyle.

Exclusion Criteria:

* Subjects with any Axis I disorder other than SAD (e.g., post-traumatic stress disorder, obsessive compulsive disorder, panic disorder) within 24 weeks of the Baseline visit. Subjects with co-morbid Major Depressive Disorder (MDD), Generalized Anxiety Disorder (GAD), dysthymia, or specific phobias will be allowed if SAD is the primary disorder in terms of clinical severity, as determined by the investigator.
* Subjects with any history or complication of schizophrenia or bipolar disorder.
* Subjects with a complication of body dysmorphic disorder.
* Substance use disorder, as defined by DSM-5 criteria, within 24 weeks of the Baseline visit.
* Subjects who are currently pregnant, lactating, or of childbearing potential and not able and willing to practice an effective method of contraception for the duration of the trial and at least 4 weeks after the final study visit.
* Subjects scoring >2 on item #3 of the HAM-D at Baseline, or who, in the opinion of the PI, are at a clinically significant risk for suicide.
* Significant risk for suicidal behavior during the course of study participation, in the opinion of the investigator, or recent (within the last 6 months prior to screening) suicidal behavior defined as scoring "yes" on items 4 or 5 in the Suicidal Ideation section of the Columbia-Suicide Severity Rating Scale (C-SSRS) at Screening or Baseline, or any suicide attempt within the 6 months prior to screening.
* Systolic blood pressure ≥165 and/or diastolic blood pressure ≥95, as measured at Screening and Baseline visits.
* Positive Urine Drug Screen at the Baseline visit, unless due to prescribed medication.
* Any current unstable and/or clinically significant medical condition, based on history or as evidenced in screening laboratory or ECG assessments.
* Current diagnosis of Diabetes Mellitus (type 1 or 2).
* Current diagnosis or past history of significant cardiovascular disease.
* Screening laboratory results showing: transaminases (ALT or AST) greater than 2 times the upper limit of normal (ULN) at screening, absolute neutrophil count (ANC) < 1000 at screening, or active Hepatitis B or Hepatitis C.
* Subjects with a history or complication of cancer or malignant tumor not in remission for at least 5 years. Basal cell skin cancers are not exclusionary.
* Any history of seizure or seizure disorder, with the exception of a single childhood febrile seizure.
* Subjects for whom cariprazine is contraindicated.
* Subjects receiving fluoxetine within 28 days of the Baseline visit.
* Subjects receiving Monoamine Oxidase Inhibitors (MAOIs) within 14 days of the Baseline visit.
* Subjects receiving any other psychotropics (including but not limited to: gabapentin, pregabalin, antipsychotics, Selective serotonin reuptake inhibitors (SSRIs), Serotonin and norepinephrine reuptake inhibitors (SNRIs), benzodiazepines, and sedative hypnotics other than zolpidem) within 14 days of the Baseline visit. Zolpidem (Ambien®) taken as needed (PRN) is allowed for insomnia if not taken more than 3 times per week.
* Subjects who started psychotherapy or Cognitive Behavioral Therapy (CBT) within 24 weeks of the Baseline visit, except for supportive psychotherapy. Subjects who have been receiving psychotherapy or CBT for more than 24 weeks prior to the Baseline visit are eligible provided that the therapy continues at the same frequency for the duration of the trial.
* Subjects receiving electro-convulsive therapy (ECT) within 12 weeks of the Baseline visit.
* Treatment refractory SAD, defined for this study as: subjects who have a history of two or more failed treatment trials with an FDA-approved SAD treatment, whereby a treatment trial is defined as a period of at least 6 weeks during which the subject received an adequate dosage of the SAD treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Change in LSAS Score | 12 Weeks or LOCF
  The primary outcome measure is the change in the Liebowitz Social Anxiety Score from Baseline to study endpoint (Week 12 or Last Observation Carried Forward (LOCF))

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Liebowitz, MD, Principal Investigator — Managing Director
Locations (1):
- The Medical Research Network, LLC, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No